CLINICAL TRIAL: NCT04941222
Title: Cost-utility Analysis of the Use of the Paro Robotic Seal by Elderly Patients With Moderate or Severe Cognitive Disorders in Institutions: a Randomised Study.
Acronym: PEPINO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of recruitment
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHD187-19
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment
Keywords: PARO; non-pharmacological intervention; economic evaluation; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With robotic seal "PARO" (Experimental): The robot will be made available to the patient by the caregiver in charge of the patient for 5 minutes before a toilet and for the duration of the treatment (about 10 minutes), twice a week for 16 weeks.
  Interventions: Other: With robotic seal "PARO"
- Without robotic seal "PARO" (No Intervention): The care of the patient during the toilet will be carried out according to the modalities currently in use in the facility.

INTERVENTIONS:
Other: With robotic seal "PARO" — The PARO robot will be made available to the patient by the caregiver in charge of the patient for 5mn before a toilet and during the duration of the care (about 10mn), at the frequency of twice a week for 16 weeks
  Arms: With robotic seal "PARO"

SUMMARY:
Many residents from establishments for dependent elderly people (EHPAD) have memory disorders with behavioural problems such as agitation, aggression and anxiety, which make it difficult to assist them on a daily basis.

Studies have proven the beneficial effect of the therapeutic seal robot PARO® in behavioural disorders. The present project aims to complement these data with a medico-economic study. At present, the only study of this type has been carried out in Australia, and is not transposable to France.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years of age
* With moderate or severe neurocognitive disorders of any etiology (Mini Mental State Examination (MMSE) less than or equal to 20, or not feasible)
* Resident in EHPAD (establishment for dependent elderly people) or USLD (long-term care unit ) in permanent accommodation for more than 1 month at inclusion

Exclusion Criteria:

* Patient with presumed life expectancy of less than 3 months
* Mini Mental State Examination (MMSE) not feasible for any reason other than cognitive impairment (e.g. stroke aphasia), without dementia
* Known carrier of multi-drug resistant bacteria
* Carrier of Pace-maker (precautionary advice from manufacturer)
* Refusal to participate to the study (trusted person, guardian or curator or patient depending on the patient's mental state)
* Patient under court protection
* Prior inclusion in an interventional study that may alter the interpretation of the results of the analysis
* Patient not affiliated to a social security system or beneficiary of such a system

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Incremental cost-utility ratio | 16 weeks after implementation of toilets with/without PARO
  Incremental cost-utility ratio (cost/QALY) from a societal perspective and a time horizon of 16 weeks of the use of the PARO robot

CONTACTS AND LOCATIONS:
Overall Officials: stéphanie CHENEAU, Principal Investigator — CHD Vendée
Locations (1):
- CHD Vendee, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No